# Postpregnancy Family Planning Choices in Public and Private Sectors in Kenya and Indonesia (PPFP Choices)

## **Informed Consent Form**

Jhpiego

Unique Protocol ID: IRB00007462

September 14, 2017

Uploaded to Clinicaltrials.gov on November 2, 2017



Approval Date: September 14, 2017 Approved Consent Version No.: 1 PI Name: Elaine Charurat IRB No. 00007462

Study Title: Postpregnancy Family Planning Choices in the Public and Private Sectors in Kenya and

Indonesia.

Study Tools: Kenya ANC Client Interview Consent

#### INFORMED CONSENT DOCUMENT

## **Kenya ANC Client Interview**

# What you should know about this study

- You are being asked to join a research study.
- This consent form explains the research study and your part in the study.
- Please read it carefully and take as much time as you need.
- You are a volunteer. You can choose not to take part and if you join, you may quit at any time. There will be no penalty if you decide to quit the study.

#### **Purpose of research project**

This research is being done to understand immediate postpartum family planning in your community and *you* are one of the experts on this topic. The information you give me will help my team develop/improve programs to help others. By talking to pregnant women and others in the community, we hope to learn how to change health services so more women want and are able to get health services when they need them.

## Why you are being asked to participate

You are being asked to participate because you are currently more than 28 weeks pregnant and have received antenatal care at a study facility. We want to talk to women in your community who will have a baby soon so we can learn what services they need, what services they have already received and how to make services better.

#### **Procedures**

If you join this study, we will ask you to do the following things:

- Meet with an interviewer up to three times, (during antenatal care visit, within 2 days of giving birth (while at the healthcare facility immediately prior to discharge), and 6 months after giving birth), for between 30-45 minutes each time.
- Discuss what you know about postpartum family planning and what your postpartum family planning needs are
- Discuss what information your doctor or other health care provider has given you about postpartum family planning
- Discuss what keeps you and others from using postpartum family planning services
- Talk about how decisions to use postpartum family planning services are made in your family and in your community
- Discuss how postpartum family planning services could be changed to make them better and easier for you to use



Approval Date: September 14, 2017 Approved Consent Version No.: 1 PI Name: Elaine Charurat IRB No. 00007462

Study Title: Postpregnancy Family Planning Choices in the Public and Private Sectors in Kenya and

Indonesia.

Study Tools: Kenya ANC Client Interview Consent

#### Risks/discomforts

You may find it uncomfortable to talk with others in your community about postpartum family planning. You can choose not to answer any question that makes you feel uncomfortable. You can leave the discussions at any time if you feel uncomfortable or for any other reason.

#### **Benefits**

There is no direct benefit to you from being in this study. However, this study is designed to obtain information to improve access to postpartum family planning. This may in turn reduce morbidity and mortality of mothers and children in the long term.

## **Payment**

There is no payment for being in this study.

## Protecting data confidentiality

All research projects carry some risk that information about you may become known to people outside of a study. We will collect personal identifiers at study enrollment to allow adequate follow-up of participants throughout the study period. We will require your name, telephone number, and secondary telephone number to ensure minimum loss to attrition during the follow-up period. After data collection is complete and there is no further need for personal identifiers, we will transform the data into a de-identified format and delete the personal identifiers within three months. To protect your information in this study, we will store your responses in a locked cabinet so that only those working in the study can read them.

## Protecting subject privacy during data collection

We will hold the interview in a private space. All answers shared with the data collector will be kept confidential.

## Who do you call if you have questions or problems?

Call the local investigator, if you have questions or complaints.

Kenya: Paul Nyachae, Project Technical Advisor, +254.200.371.882

Call or contact the local IRB if you have questions about your rights as a study participant.
 Contact the local IRB if you feel you have not been treated fairly or if you have other concerns. The local IRB contact information is:

Kenya:

KEMRI Scientific Ethics Review Committee

P.O Box 54840-00200, Nairobi;

Phone: 020-2722541, 0722205901, 0733400003;



Approval Date: September 14, 2017 Approved Consent Version No.: 1 PI Name: Elaine Charurat IRB No. 00007462

Study Title: Postpregnancy Family Planning Choices in the Public and Private Sectors in Kenya and Indonesia.

Study Tools: Kenya ANC Client Interview Consent

## What does your permission mean?

Your permission means:

- You have been informed about this study's purpose, procedures, possible benefits and risks.
- You have been given the chance to ask questions.
- You have voluntarily agreed to be in this study.

| Individual consents to participate in study | | |
|---|---|---|
| Print name of Person Obtaining Consent | Signature of Person Obtaining Consent | –<br>Date |
| Print name of Participant Date | Signature or mark of Participant | _ |
| Give one copy to the p | articipant and keep one copy in study reco | rds |